CLINICAL TRIAL: NCT05107843
Title: Integrated Clinical-radiological Analysis of Hypoxia Markers in Pediatric Osteosarcomas - Single-center Pilot Study of 32 Patients
Brief Title: Integrated Clinical-radiological Analysis of Hypoxia Markers in Pediatric Osteosarcomas
Acronym: SARCOMAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7715
Record Dates: First submitted 2021-10-05; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Osteosarcoma in Children
Keywords: Osteosarcoma; Necrosis; Immunohistochemical markers of hypoxia; Hypoxia; Chemotherapy; Metastasis
MeSH Terms: conditions — Osteosarcoma; Necrosis; Hypoxia; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this pilot study is therefore to retrospectively measure the volume and percentage of necrosis on diagnostic MRI in T1 sequence and in parallel to study the expression of immunohistochemical markers of hypoxia (HIF-1α, CAIX , HIF-2α, pS6, phosphomTor, CD163 and CD68) on diagnostic biopsies of high-grade osteosarcomas from 2007 to 2018 in the Strasbourg center, focusing on the pediatric population. The investigators will systematically carry out a correlation analysis between these different parameters and with the clinical data of these same patients (response to chemotherapy, presence of metastases or not and overall and recurrence-free survival). This will eventually make it possible to highlight new prognostic markers at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≤ 20 years at diagnosis
* Subject having been treated for osteosarcoma in the OS2006 protocol or treated according to
* Supported at Strasbourg University Hospitals between 05/01/2007 and 10/31/2018
* Availability of its diagnostic tumor material stored in paraffin
* having an MRI diagnostic evaluation comprising the injected T1 sequences necessary for the analysis of the volume / necrotic proportion.

Exclusion Criteria:

* Opposition of the patient (or his legal representatives if he is a minor) to participate in the study
* Diagnosis other than osteosarcoma
* Biological tissue from a patient who does not meet all the inclusion criteria
* Patient under legal protection
* Patient under guardianship or guardianship

Ages: 1 Year to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subject ≤ 20 years having been treated for osteosarcoma in the OS2006 protocol or treated according to.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Retropsective study of pediatric osteosarcomas | Files analysed retrospectively from January 01, 2007 to December 31, 2018 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Natacha ENTZ-WERLE, MD, PhD, Principal Investigator — Service Pédiatrie Onco-hématologie - Pédiatrie III - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service Pédiatrie Onco-hématologie - Pédiatrie III - Hôpitaux Universitaires de Strasbourg, Strasbourg, France